CLINICAL TRIAL: NCT00730132
Title: Observational Study of Approaches to Lipid-lowering Therapy in Russian Patients With Coronary Heart Disease (<<Treat to Goal>>)
Brief Title: Observational Study of Approaches to Lipid-Lowering Therapy in Russian Patients With Coronary Heart Disease <<Treat to Goal>> (Study P05464)
Status: Completed | Type: Observational
Sponsor: Organon and Co (Industry)
Responsible Party: Sponsor
Other Study IDs: P05464
Record Dates: First submitted 2008-07-25; First posted 2008-08-08 (Estimated); Results first posted 2010-10-11 (Estimated); Last update posted 2022-02-09 (Actual); Status verified 2022-02

CONDITIONS: Coronary Heart Disease; Hypercholesterolemia
MeSH Terms: conditions — Coronary Disease; Hypercholesterolemia | interventions — Ezetimibe; Hydroxymethylglutaryl-CoA Reductase Inhibitors

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- New Statin: Group 1 - Patients with established diagnosis of CHD and hypercholesterolemia who did not achieve the target values for TC and LDL-C with existing statin therapy (atorvastatin, fluvastatin, lovastatin, pravastatin, rosuvastatin, simvastatin) whose lipid-lowering therapy was modified by transition to a new statin treatment
  Interventions: Drug: Statin
- Statin Dose Titration: Group 2 - Patients with established diagnosis of CHD and hypercholesterolemia who did not achieve the target values for TC and LDL-C with existing statin therapy (atorvastatin, fluvastatin, lovastatin, pravastatin, rosuvastatin, simvastatin) whose lipid-lowering therapy was modified by increasing the dose of ongoing statin treatment
  Interventions: Drug: Statin
- Ezetimibe added to existing statin: Group 3 - Patients with established diagnosis of CHD and hypercholesterolemia who did not achieve the target values for TC and LDL-C with existing statin therapy (atorvastatin, fluvastatin, lovastatin, pravastatin, rosuvastatin, simvastatin) and whose lipid-lowering therapy was modified by the addition of ezetimibe to ongoing statin treatment
  Interventions: Drug: Ezetimibe

INTERVENTIONS:
Drug: Ezetimibe — Dosage determined by the investigator based on standard and applicable routine clinical practice for CHD and hypercholesterolemia patients
  Other Names: SCH 58235; Ezetrol
  Groups: Ezetimibe added to existing statin
Drug: Statin — Statin titration for the Statin Dose Titration group, and new statin treatment and dosage for the New Statin group, determined by the investigator based on standard and applicable routine clinical practice for CHD and hypercholesterolemia patients
  Groups: New Statin; Statin Dose Titration

SUMMARY:
This study is being performed to evaluate what variants of lipid-lowering therapy are used in Russian clinical practice in coronary heart disease (CHD) patients with hypercholesterolemia in whom the initial statin therapy did not achieve low density lipoprotein-cholesterol (LDL-C) goals. Additionally, the efficacy and safety of all variants of modified lipid-lowering therapy are to be evaluated.

DETAILED DESCRIPTION:
Given the observational nature of this study and that the assessment of a specific hypothesis is not foreseen, statistical assumption is not planned and the sample size calculation was not performed.

Taking into consideration the available data on the established safety profile of the therapy with statins and combination of ezetimibe with statins it has been suggested that a sample size of 750 patients will be sufficient to identify adverse events profile.

The treatment effects will be characterized by descriptive and frequency parameters.

ELIGIBILITY:
Inclusion Criteria:

* Male and Female, from 18 to 75 years old;
* Established diagnosis of CHD;
* Previous (at least, within 1 month before inclusion in the present study) treatment with statin;
* Levels of plasma TC and LDL-C above the recommended target values

(TC> 4.5 mmol\L; LDL-C> 2.5 mmol/L);

* The written informed consent signed prior to the start of participation in the study.

Exclusion Criteria:

* Contraindications for statin and ezetimibe (Ezetrol) administration in accordance with local Russian Federation medical instructions.
* Patients refused to participate in the study and/or did not sign informed consent form.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with established diagnosis of coronary heart disease (CHD) and hypercholesterolemia who did not achieve the target values for total cholesterol (TC) and low density lipoprotein-C (LDL-C) with existing statin therapy
Sampling Method: Non-Probability Sample
Enrollment: 712 (Actual)
Dates: Start 2008-01; Primary Completion 2009-08 (Actual); Study Completion 2009-08 (Actual)

RESULTS

PARTICIPANT FLOW:
Groups:
- Enrolled Patients: Patients with established diagnosis of CHD and hypercholesterolemia who did not achieve the target values for TC and LDL-C with existing statin therapy and who consented to enroll in this observational study, allowing collection of data regarding change in treatment, and treatment efficacy and safety.
Period: Overall Study
Arm/Group | Enrolled Patients
Started | 712
Completed | 557
Not Completed | 155
Not completed — Protocol Violation | 154
Not completed — Death | 1

BASELINE CHARACTERISTICS:
Arm/Group | Enrolled Patients
Number analyzed (Participants) | 712
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.57 (9.367)
Sex/Gender, Customized [Number; unit: participants]
  Female | 324
  Male | 386
  Not Reported | 2
Region of Enrollment [Number; unit: participants]
  Russian Federation | 712

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Patients Receiving Each Variant of Modified Lipid-lowering Therapy: Statin Dose Titration, Administration of a New Statin, Administration of a Ezetimibe in Addition to a Current Statin.
Description: Statins included: 1. statin dose (atorvastatin, fluvastatin, rosuvastatin, simvastatin) titration . 2. shift to a (atorvastatin, fluvastatin, lovastatin, pravastatin, rosuvastin, simvastatin) different statin . 3. Ezetimibe added to existing statin (atorvastatin, lovastatin, rosuvastatin, simvastatin).
Time Frame: During the study
Population: The efficacy analysis set (n=557) included all enrolled subjects, by treatment (after treatment modification), who received at least one dose of the modified lipid-lowering treatment and for whom no protocol violations were recorded. One subject each from ezetimibe added to existing statin and new statin group were excluded (missing data)
Measure: Number; unit: Percentage of patients
Groups:
- All Participants Analyzed: Patients with established diagnosis of CHD and hypercholesterolemia who did not achieve the target values for TC and LDL-C. A participant was included in the study in case the lipid lowering therapy was modified in one of the following options: 1- statin dose (atorvastatin, fluvastatin, lovastatin, pravastatin, rosuvastatin, simvastatin) titration, 2- administration of a new statin (atorvastatin, fluvastatin, lovastatin, pravastatin, rosuvastatin, simvastatin), 3- administration of ezetimibe in addition to current statin (atorvastatin, fluvastatin, lovastatin, pravastatin, rosuvastatin, simvastatin) therapy.
Arm/Group | All Participants Analyzed
Number analyzed (Participants) | 557
Percentage of patients
  Statin dose titration | 32.1
  New statin administered | 42.4
  Ezetimibe added on to existing statin | 25.5

2. Primary Outcome: Percentage of Patients Per Group Who Reach Goal for Total Cholesterol (TC) (< 4.5 mmol/L) According to All-Russian Scientific Cardiologists Society (ARSCS) Recommendations by End of Observation
Description: Statins included in this outcome measure included: 1. statin dose (atorvastatin, fluvastatin, rosuvastatin, simvastatin) titration. 2. shift to a different (atorvastatin, fluvastatin, lovastatin, pravastatin, rosuvastin, simvastatin) statin . 3. Ezetimibe added to existing statin (atorvastatin, lovastatin, rosuvastatin, simvastatin).
Time Frame: Visit 2 (Month 2, end of observation)
Population: The efficacy analysis set (n=557) included all enrolled subjects, by treatment (after treatment modification), who received at least one dose of the modified lipid-lowering treatment and for whom no protocol deviations were recorded. One subject each from the Ezetimibe and New Statin groups were excluded from this analysis due to missing data.
Measure: Number; unit: Percentage of patients
Groups:
- Ezetimibe Added to Existing Statin: Patients with established diagnosis of CHD and hypercholesterolemia who did not achieve the target values for TC and LDL-C with existing statin therapy (atorvastatin, fluvastatin, lovastatin, pravastatin, rosuvastatin, simvastatin) and whose lipid-lowering therapy was modified by the addition of ezetimibe to ongoing statin
- Statin Dose Titration: Patients with established diagnosis of CHD and hypercholesterolemia who did not achieve the target values for TC and LDL-C with existing statin therapy (atorvastatin, fluvastatin, lovastatin, pravastatin, rosuvastatin, simvastatin) and whose lipid-lowering therapy was modified by increasing the dose of ongoing statin therapy
- New Statin: Patients with established diagnosis of CHD and hypercholesterolemia who did not achieve the target values for TC and LDL-C with existing statin therapy (atorvastatin, fluvastatin, lovastatin, pravastatin, rosuvastatin, simvastatin) and whose lipid-lowering therapy was modified by transition to a new statin therapy
Arm/Group | Ezetimibe Added to Existing Statin | Statin Dose Titration | New Statin
Number analyzed (Participants) | 141 | 179 | 235
Percentage of patients | 50.4 | 33.5 | 37.4
Statistical Analysis 1: Comparison: Ezetimibe Added to Existing Statin vs Statin Dose Titration vs New Statin; Significance of the differences in the number of patients per group who achieved goal TC levels on Visit 2; Test type: Superiority or Other; p = 0.007, Pearson Chi-Square

3. Primary Outcome: Percentage of Patients Per Group Who Reached Goal for Low Density Lipoprotein (LDL-C) (< 2.6 mmol/L) According to ARSCS Recommendations by End of Observation
Time Frame: Visit 2 (Month 2, end of observation)
Population: The efficacy analysis set (n=557) included all enrolled subjects, by treatment (after treatment modification), who received at least one dose of the modified lipid-lowering treatment and for whom no protocol deviations were recorded.
Measure: Number; unit: Percentage of patients
Arm/Group | Ezetimibe Added to Existing Statin | Statin Dose Titration | New Statin
Number analyzed (Participants) | 142 | 179 | 235
Percentage of patients | 42.3 | 26.3 | 33.9
Statistical Analysis 1: Comparison: Ezetimibe Added to Existing Statin vs Statin Dose Titration vs New Statin; Significance of paired changes in the number of patients who achieved LDL-C target levels on Visit 2, for each treatment group comparison; Test type: Superiority or Other; p < 0.001, McNemar — Chi square, continuity corrected. Asymptotic significance

4. Primary Outcome: Percentage of Relative Change of Total Cholesterol (TC) Level Measured on Visit 2 Compared With the Baseline (Visit 1) in Each of the Three Therapy Groups
Time Frame: Visit 2 (Month 2, end of observation) and Visit 1 (Day 0, baseline)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Ezetimibe Added to Existing Statin | Statin Dose Titration | New Statin
Number analyzed (Participants) | 141 | 179 | 235
mmol/L | 25.76 (12.306) | 20.01 (15.662) | 22.82 (14.035)
Statistical Analysis 1: Comparison: Ezetimibe Added to Existing Statin; Descriptive statistics of relative (%) change in TC levels from Baseline at Visit 2; Test type: Superiority or Other; Mean Difference (Final Values) = 25.7570, Standard Deviation 12.30606
Statistical Analysis 2: Comparison: Statin Dose Titration; Descriptive statistics of relative (%) change in TC from baseline at Visit 2; Test type: Superiority or Other; Mean Difference (Final Values) = 20.00, Standard Deviation 15.662
Statistical Analysis 3: Comparison: New Statin; Descriptive statistics of relative (%) change in TC from baseline at Visit 2; Test type: Superiority or Other; Mean Difference (Final Values) = 22.8181, Standard Deviation 14.03545
Statistical Analysis 4: Comparison: Statin Dose Titration vs New Statin; Statin Dose Titration compared to New Statin; Test type: Superiority or Other; p = .143, Games-Howell; Mean Difference (Final Values) = -2.80928, 95% CI 2-sided [-6.3070 to .6884], Standard Error of Mean 1.48621
Statistical Analysis 5: Comparison: Ezetimibe Added to Existing Statin vs Statin Dose Titration; Statin Dose Titration compared to Ezetimbe; Test type: Superiority or Other; p = .001, Games-Howell; Mean Difference (Final Values) = -5.74811, 95% CI 2-sided [-9.4298 to -2.0664], Standard Error of Mean 1.56351
Statistical Analysis 6: Comparison: Ezetimibe Added to Existing Statin vs New Statin; New Statin compared to Ezetimibe; Test type: Superiority or Other; p = .086, Games-Howell; Mean Difference (Final Values) = -2.93883, 95% CI 2-sided [-6.1948 to .3171], Standard Error of Mean 1.38286

5. Primary Outcome: Percentage of Relative Change of LDL-C Level Measured on Visit 2 Compared With the Baseline (Visit 1) in Each of the Three Therapy Groups
Time Frame: Visit 2 (Month 2, end of observation) and Visit 1 (Day 0, baseline)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Ezetimibe Added to Existing Statin | Statin Dose Titration | New Statin
Number analyzed (Participants) | 142 | 179 | 235
mmol/L | 32.06 (15.590) | 26.81 (19.852) | 28.24 (20.787)
Statistical Analysis 1: Comparison: Statin Dose Titration; Descriptive statistics of relative (%) change in LDL-C levels by the end of the study (Visit 2) compared to Baseline (Visit 1); Test type: Superiority or Other; Mean Difference (Final Values) = 26.8174, Standard Deviation 19.85205
Statistical Analysis 2: Comparison: New Statin; [analysis description as in outcome 5, analysis 1]; Test type: Superiority or Other; Mean Difference (Final Values) = 28.2488, Standard Deviation 20.78727
Statistical Analysis 3: Comparison: Ezetimibe Added to Existing Statin; [analysis description as in outcome 5, analysis 1]; Test type: Superiority or Other; Mean Difference (Final Values) = 32.0665, Standard Deviation 15.59010
Statistical Analysis 4: Comparison: Statin Dose Titration vs New Statin; Statin Dose Titration compared to New Statin; Test type: Superiority or Other; p = .756, Games-Howell; Mean Difference (Final Values) = -1.43138, 95% CI 2-sided [-6.1604 to 3.2977], Standard Error of Mean 2.01009
Statistical Analysis 5: Comparison: Ezetimibe Added to Existing Statin vs Statin Dose Titration; Statin Dose Titration compared to Ezetimibe; Test type: Superiority or Other; p = .023, Games-Howell; Mean Difference (Final Values) = -5.24911, 95% CI 2-sided [-9.9072 to -.5910], Standard Error of Mean 1.97821
Statistical Analysis 6: Comparison: Ezetimibe Added to Existing Statin vs New Statin; New Statin compared to Ezetimibe; Test type: Superiority or Other; p = .107, Games-Howell; Mean Difference (Final Values) = -3.81773, 95% CI 2-sided [-8.2523 to .6169], Standard Error of Mean 1.88425

ADVERSE EVENTS:
Description: Adverse Events (AEs) and Serious Adverse Events (SAEs) are represented for all treatment subjects (n=712) not by treatment group because in this observational study the three treatment group populations cannot be clearly identified for a substantial number of subjects.
Arm/Group | Enrolled Patients
Serious Adverse Events (participants affected / at risk) | 3/712
Other Adverse Events (participants affected / at risk) | 0/712
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Enrolled Patients (N=712)
Cardiac asthma (Cardiac disorders) | 1 (1)
Cardiac failure congestive (Cardiac disorders) | 1 (1)
Coronary artery disease (Cardiac disorders) | 1 (1)
Gastric hemorrhage (Gastrointestinal disorders) | 1 (1)
Hypotonia (Nervous system disorders) | 1 (1)
Vascular graft (Surgical and medical procedures) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A disclosure agreement restricts the rights on publications within 5 years after the document is signed off. The Clinical Trial Agreement restricts the rights on publication within 5 years after the trial completion.